CLINICAL TRIAL: NCT01326689
Title: Phase III Study of KW-2246 (A Double Blind Study of KW-2246 Compared to Placebo for Breakthrough Pain Episodes in Cancer Patients)
Brief Title: A Comparative Study of KW-2246
Acronym: 2246-004
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2246-004
Record Dates: First submitted 2011-03-30; First posted 2011-03-31 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Cancer Related Pain (Breakthrough Pain)
MeSH Terms: conditions — Cancer Pain; Breakthrough Pain

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- KW-2246 (Experimental)
  Interventions: Drug: KW-2246
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KW-2246 — Rescue medication at an optimal dose, which is determined by dose titration
  Arms: KW-2246
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a placebo-controlled, double blind, comparative study to evaluate the efficacy and safety of KW-2246 as rescue medication at an optimal dose, which is determined by dose titration in treating breakthrough pain episodes in adult cancer patients receiving strong opioid analgesic on a fixed-schedule as well as rescue medication for breakthrough pain.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Have been treated with opioid analgesic on a fixed-schedule at a stable daily dose
* Receiving at least 1 but not more than 4 doses of rescue medication per day in average and whose pain is controlled
* ECOG PS =< 3

Exclusion Criteria:

* Currently suffered from intolerable opioid-specific adverse reactions due to opioid analgesics
* Severe respiratory dysfunction
* Asthma
* Severe bradyarrhythmia
* Severe hepatic function disorder
* Severe renal function disorder
* Severe psychoneurotic disorder
* Susceptibility to respiratory depression due to such conditions as increased intracranial pressure, head injury or brain tumor

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Pain intensity difference | 30 minutes after each dose
  Pain scores on the visual analog scale

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo, Japan

REFERENCES:
- [Derived] Shimoyama N, Gomyo I, Katakami N, Okada M, Yukitoshi N, Ohta E, Shimoyama M. Efficacy and safety of sublingual fentanyl orally disintegrating tablet at doses determined by titration for the treatment of breakthrough pain in Japanese cancer patients: a multicenter, randomized, placebo-controlled, double-blind phase III trial. Int J Clin Oncol. 2015 Feb;20(1):198-206. doi: 10.1007/s10147-014-0697-z. Epub 2014 May 20. PMID 24839047